CLINICAL TRIAL: NCT00291070
Title: A Double Blind, Randomized Placebo Controlled Clinical Trial Examining the Effects of L-Theanine (Suntheanine®) in Male Child Subjects With Attention Deficit Hyperactivity Disorder
Brief Title: Effects of L-Theanine in Boys With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Michael Lyon, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C04-0605
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; attention; insomnia; hyperactivity; anxiety
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Initiation and Maintenance Disorders; Spasm; Anxiety Disorders | interventions — theanine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: L-theanine — This study will examine the effects of L-theanine (an amino acid found in green tea) on the behavior, cognitive performance and sleep quality of boys with ADHD.

SUMMARY:
This study will examine the effects of L-theanine (an amino acid found in green tea) on the behavior, cognitive performance and sleep quality of boys with ADHD.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of attention deficit hyperactivity disorder (ADHD)

Exclusion Criteria:

-

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Cognitive performance

SECONDARY OUTCOMES:
Sleep quality, hyperactive behaviors, anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Lyon, Principal Investigator — University of British Columbia
Locations (1):
- Canadian Center for Functional Medicine, Coquitlam, British Columbia, Canada